CLINICAL TRIAL: NCT02696044
Title: Treatment of Mitochondrial Dysfunction in Rett Syndrome With Triheptanoin: An Open-label, 10-subject Clinical Trial of UX007 (Triheptanoin) in the Treatment of Mitochondrial Dysfunction in Participants With Rett Syndrome, Dyskinesia, and Epilepsy
Brief Title: Treatment of Mitochondrial Dysfunction in Rett Syndrome With Triheptanoin
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Center for Rare Neurological Diseases, Norcross, GA (Other)
Collaborators: Ultragenyx Pharmaceutical Inc (Industry); Rett Syndrome Research Trust (Other)
Responsible Party: Principal Investigator, Daniel C. Tarquinio, Managing Director, Center for Rare Neurological Diseases, Norcross, GA
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00085194
Record Dates: First submitted 2016-02-25; First posted 2016-03-02 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Rett Syndrome
Keywords: Gastrointestinal Disorders
MeSH Terms: conditions — Rett Syndrome; Gastrointestinal Diseases | interventions — triheptanoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Participants aged 0 months to 3 years (Experimental): Participants will receive 4 grams of triheptanoin per kilogram of body weight daily.
  Interventions: Drug: triheptanoin
- Participants aged 4 to 6 years (Experimental): Participants will receive 3 grams of triheptanoin per kilogram of body weight daily.
  Interventions: Drug: triheptanoin
- Participants aged 7 to 9 years (Experimental): Participants will receive 2.5 grams of triheptanoin per kilogram of body weight daily.
  Interventions: Drug: triheptanoin
- Participants aged 10 to 14 years (Experimental): Participants will receive 2 grams of triheptanoin per kilogram of body weight daily.
  Interventions: Drug: triheptanoin
- Participants aged 15 to 20 years (Experimental): Participants will receive 1.5 grams of triheptanoin per kilogram of body weight daily.
  Interventions: Drug: triheptanoin
- Participants aged 21 years and older (Experimental): Participants will receive 1.2 grams of triheptanoin per kilogram of body weight daily.
  Interventions: Drug: triheptanoin

INTERVENTIONS:
Drug: triheptanoin — Participants will begin a 2 week dose titration period to achieve study drug treatment comprising of 1-4 grams per kilogram of body weight (g/kg) daily depending on age. The age-related target dose will be mixed with food or formula and administered orally or by gastronomy tube. The total daily dose can be divided into 4 equal doses taken 4 times daily. Participants will maintain the age dependent dose treatment at the 1-4 g/kg daily for four months.

SUMMARY:
The aim of this study is to evaluate the safety and tolerability of triheptanoin in participants with Rett syndrome using laboratory values, electrocardiogram, rate of adverse events (AE), and physical exam.This study also seeks to evaluate the efficacy of UX007 (triheptanoin) in improving overall seizure frequency and dystonia.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the safety and tolerability of triheptanoin in participants with Rett syndrome using laboratory values, electrocardiogram, rate of adverse events (AE), and physical exam. This study also seeks to evaluate the efficacy of UX007 (triheptanoin) in improving overall seizure frequency, dystonia severity, and quality of life. Participants who are eligible will take triheptanoin daily. Participation in the primary arm of this study will last up to 8.5 months, with an optional 36 month extension.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Classic Rett syndrome as defined by the clinical consensus criteria
* Presence of a MECP2 mutation
* Post-regression stage of development, defined as greater than 6 months since the last loss of hand use or verbal language
* Average of at least 4 observable seizures (generalized or partial-onset [Generalized Tonic-Clonic, Generalized Tonic, Generalized Clonic, Generalized Atonic, Partial/Focal with Secondary Generalization, Myoclonic, Myoclonic Atonic, Myoclonic Tonic, Complex Partial/Focal, and Simple Partial/Focal Motor) in one month prior to the study by caregiver report or presence of dystonia on average at least four times in one month prior to the study in at least one body region rated as at least "mild" by caregiver report
* Use of at least one anti-seizure medication at screening visit
* At screening visit, managed on four or fewer concomitant anti-seizure medications that must have been stable in dose at least one month prior to the beginning of screening and anticipated to remain stable in dose through the end of the 8.5 month trial period
* Legally authorized caregiver must be willing to give written informed consent after the nature of the study has been explained, and prior to any research-related procedures
* Caregiver and participant must, in the opinion of the investigator, be willing and able to complete all aspects of the study, comply with accurate completion of the seizure and dystonia diaries, and be likely to complete the four month treatment period

Exclusion Criteria:

* Markedly abnormal metabolic screening laboratory testing (e.g., serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels exceeding 2X the upper limit of normal)
* Any known hypersensitivity to triheptanoin that, in the judgment of the investigator, places the subject at increased risk for adverse effects
* Prior use of triheptanoin within 1 month prior to screening
* Participants or caregivers who are unwilling or unable to discontinue use of a prohibited medication or other substance that may confound study objectives
* Use of any other investigational product, including drugs or supplements within 1 month prior to Screening, or at any time during the study
* Has a condition of such severity and acuity, in the opinion of the investigator, that it warrants immediate surgical intervention or other treatment
* Has a concurrent disease or condition, or laboratory abnormality that, in the view of the investigator, places the subject at high risk of poor treatment compliance or of not completing the study, or would interfere with study participation or introduces additional safety concerns (e.g., diabetes mellitus)
* Pregnant or nursing women

Min Age: 2 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-06; Primary Completion 2021-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Seizure Frequency | Visit 2, Visit 7 (Up to 4 months)
  The number of observable seizures recorded via caregiver-reported diary between Visit 2 and Visit 7 of treatment.
Change in Dystonia frequency | Visit 2, Visit 7 (Up to 4 months)
  The frequency of dystonic posturing present in each limb recorded via caregiver-reported diary on each day of treatment between Visit 2 and Visit 7 of treatment.

SECONDARY OUTCOMES:
Change in Dystonia Severity | Visit 1, Visit 7 (Up to 4 months)
  The percentage of participants with a median improvement of at least 50% in their degree of dystonia severity in all body regions averaged together from the baseline period to the end of the treatment period.
Change in Burke-Fahn-Marsden Dystonia Rating Scale (BFM) Score | Visit 1, Visit 9 (Up to 8.5 months)
  The BFM s a 120-point rating scale used to test the severity of dystonia in 9 body regions. This scale takes into account the severity and frequency of the dystonic movements. A higher score means greater impairment.
Change in Global Dystonia Rating Scale (GDRS) Score | Visit 1, Visit 9 (Up to 8.5 months)
  The GDS rates dystonia in 14 body areas. The GDS is a Likert type scale with ratings from 0 to 10 (0 is no dystonia, 1 minimal, 5 moderate and 10 severe dystonia). A higher score represents more severe dystonia.
Change in the PROMIS Fatigue Parent Proxy Score | Visit 2, Visit 7 (Up to 4 months)
  The Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue Parent Proxy evaluates a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. Fatigue is divided into the experience of fatigue (frequency, duration, and intensity) and the impact of fatigue on physical, mental, and social activities. Scores range from 0 to 40 with a higher score indicating higher fatigue impact.
Change in the PROMIS Pain Interference Parent Proxy Score | Visit 2, Visit 7 (Up to 4 months)
  The Patient Reported Outcomes Measurement Information System (PROMIS) Pain Interference Parent Proxy measures the self-reported consequences of pain on relevant aspects of one's life. This includes the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. It assesses pain interference over the past seven days. Scores range from 0 to 40 with a higher score indicating higher pain interference.
Change in the PROMIS Peer Relations Parent Proxy Score | Visit 2, Visit 7 (Up to 4 months)
  The Patient Reported Outcomes Measurement Information System (PROMIS) Peer Relations Parent Proxy assesses the quality of relationships with friends and other acquaintances. Scores range from 0 to 28. A higher score indicates better peer relations.
Change in the PROMIS Physical Functional Mobility Parent Proxy Score | Visit 2, Visit 7 (Up to 4 months)
  The Patient Reported Outcomes Measurement Information System (PROMIS) Physical Functional Mobility Parent Proxy measures self-reported capability rather than actual performance of physical activities. This includes the functioning of one's upper extremities (dexterity), lower extremities (walking or mobility), and central regions (neck, back), as well as instrumental activities of daily living, such as running errands. Each form assesses current function rather than function over a specified time period. Scores range from 0 to 32 with a lower score indicating lower mobility.
Change in the PROMIS Physical Function Upper Extremity Parent Proxy Score | Visit 2, Visit 7 (Up to 4 months)
  The Patient Reported Outcomes Measurement Information System (PROMIS) Physical Function Upper Extremity Parent Proxy measures self-reported capability rather than actual performance of physical activities. This includes the functioning of one's upper extremities (dexterity), lower extremities (walking or mobility), and central regions (neck, back), as well as instrumental activities of daily living, such as running errands. Each form assesses current function rather than function over a specified time period. Scores range from 0 to 32 with a lower score indicating lower mobility.
Change in the PROMIS Anxiety Parent Proxy Score | Visit 2, Visit 7 (Up to 4 months)
  The Patient Reported Outcomes Measurement Information System (PROMIS) Anxiety Parent Proxys measures self-reported fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness). Anxiety is assessed over the past seven days. Scores range from 0 to 32 with a higher score indicating higher anxiety.
Change in the PROMIS Depressive Symptoms Parent Proxy Score | Visit 2, Visit 7 (Up to 4 months)
  The Patient Reported Outcomes Measurement Information System (PROMIS) Anxiety Parent Proxys assessed self-reported negative mood (sadness, guilt), views of self (selfcriticism, worthlessness), and social cognition (loneliness, interpersonal alienation), as well as decreased positive affect and engagement (loss of interest, meaning, and purpose). It assesses depression over the past seven days. Scores range from 0 to 32 with higher score indicating more depressive symptoms.
Change in Child Health Questionnaire-50 (CHQ) Score | Visit 2, Visit 7 (Up to 4 months)
  The CHQ is a self administered quality of life measure of 14 physical and psychosocial concepts and assesses a child's physical, emotional, and social well-being from the perspective of a parent or guardian.
Change in the Clinician Clinical Global Impression - Improvement Scale (CGI-S) Score | Visit 2, Visit 9 (Up to 8.5 months)
  The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the participant's illness at the time of assessment, relative to the clinician's past experience with participants who have the same diagnosis. Considering total clinical experience, a participant is assessed on severity of mental illness at the time of rating 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
Change in the Clinician Clinical Global Impression - Severity Scale Score | Visit 2, Visit 9 (Up to 8.5 months)
  The Clinical Global Impression - Improvement scale (CGI-I) is a 7 point scale that requires the clinician to assess how much the participant's illness has improved or worsened relative to a baseline state at the beginning of the intervention. and rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
Change in the Parental Clinical Global Impression of Improvement Score | Visit 2, Visit 9 (Up to 8.5 months)
  The Parental Clinical Global Impression of Improvement Scale is a 7 point scale that requires the parent/guardian to assess how much the participant's illness has improved or worsened relative to a baseline state at the beginning of the intervention. and rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
Change in Parent Top Three Concerns Visual Analog Scale Ranking | Visit 2, Visit 9 (Up to 8.5 months)
  Parents/caregivers will rank their most concerning top three symptoms associated with their child's diagnosis of Rett syndrome. Rankings range on a line scale from best to worst.
Change in the Clinical Severity Scale (CSS) Score | Visit 1, Visit 9 (Up to 8.5 months)
  The Clinical Severity Scale is a measure of onset or disease regression, growth, motor and communication skills, and disease behaviors. Measures are rated on a severity scale from 0 to 5. A higher score indicates more progressive disease.
Change in the Motor Behavioral Assessment (MBA) Score | Visit 1, Visit 9 (Up to 8.5 months)
  The MBA is a measure of onset or disease regression, growth, motor and communication skills, and disease behaviors. Measures are rated on a severity scale from 0 to 5. A higher score indicates more progressive disease.
Change in the Rett Syndrome Behavioural Questionnaire (RSBQ) Score | Visit 1, Visit 9 (Up to 8.5 months)
  The RSBQ is a self-administered questionnaire completed by caregivers. The RSBQ measures frequency of disease behaviors on a scale from 0 to 2 (0 indicating a statement is not true, 1 indicating a statement is somewhat or sometimes true, and 2 indicating a statement is very true).
Change in the Rett Syndrome Hand Apraxia Scale (RHAS) Score | Visit 1, Visit 9 (Up to 8.5 months)
  The Hand Apraxia Scale is a validated 10-item scale, with a score for a given task being 1 if it could be performed and 2 if it could not.
Change in the Rett Syndrome Gross Motor Scale (RSGMS) Score | Visit 1, Visit 9 (Up to 8.5 months)
  The RSGMS assesses the ability of subjects to sit, transfer to standing, stand, walk, side-step, turn, bend, step over obstacles, walk and run. Completion time for videotaping by parents is typically 30 45 minutes.
Change in Maximum Heart Rate as assessed by the Graded Maximal Treadmill Test | Visit 1, Visit 9 (Up to 8.5 months)
  Participants will begin walking at 3 KPH. The speed will be increased each minute by a set amount (alternating between 0.3 and 0.2 KPH). The test will continue until one of three outcomes occurs: 1) the participant indicates they would like to stop, 2) the predicted maximum heart rate (90) is reached, or the principal investigator or therapist determines the subject should no longer continue. In each possible outcome, the maximum speed achieved during the final full-minute stage will be recorded. The participant will rest, and the test will be repeated, with the goal to achieve one speed interval (0.3 or 0.2 KPH) higher than the previous test. The maximal heart rate will be recorded as the heart rate at the end of the first and second walk.
Change in Maximum Speed Acheived as assessed by the Graded Maximal Treadmill Test | Visit 1, Visit 9 (Up to 8.5 months)
  Participants will begin walking at 3 KPH. The speed will be increased each minute by a set amount (alternating between 0.3 and 0.2 KPH). The test will continue until one of three outcomes occurs: 1) the participant indicates they would like to stop, 2) the predicted maximum heart rate (90) is reached, or the principal investigator or therapist determines the subject should no longer continue. In each possible outcome, the maximum speed achieved during the final full-minute stage will be recorded.
Frequency of Epileptiform Electroencephalogram (EEG) Activity | Visit 1, Visit 7 (Up to 6.5 months)
  EEG monitoring will be performed for 24 hours with a standard 21 electrode international 10-20 protocol. Frequency of EEG activity will be measured by manual spike counting and frequency of clinical and subclinical electrographic seizures.
Seizure Activity assessed by Change in Photoplethysmographic Heart Rate | Visit 1, Visit 9 (Up to 8.5 months)
  Photoplethysmographic heart rate will be measured using the Empatica E4 watch which has a built-in algorithm for seizure prediction.
Change in Daily 3-axis accelerometry | Visit 1, Visit 9 (Up to 8.5 months)
  Accelerometry will be measured using the Empatica E4 watch which has a built-in algorithm for measuring step count.
Seizure Activity assessed by Change in Electrodermal Activity (EDA) | Visit 1, Visit 9 (Up to 8.5 months)
  Electrodermal Activity (EDA) will be measured using the Empatica E4 watch which has a built-in algorithm for seizure prediction.
Seizure Activity assessed by Change in Skin Temperature | Visit 1, Visit 9 (Up to 8.5 months)
  Skin Temperature will be measured using the Empatica E4 watch which has a built-in algorithm for seizure prediction.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Tarquinio, DO, Principal Investigator — Center for Rare Neurological Diseases
Locations (1):
- Center for Rare Neurological Diseases, Norcross, Georgia, United States

REFERENCES:
- [Derived] Hou W, Bhattacharya U, Pradana WA, Tarquinio DC. Assessment of a Clinical Trial Metric for Rett Syndrome: Critical Analysis of the Rett Syndrome Behavioural Questionnaire. Pediatr Neurol. 2020 Jun;107:48-56. doi: 10.1016/j.pediatrneurol.2020.01.009. Epub 2020 Feb 4. PMID 32165033